CLINICAL TRIAL: NCT01375582
Title: Objective Evaluation of Ocular Surface Lubricants
Brief Title: Objective Evaluation of Ocular Surface Lubricants in Two Environments
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, James V. Aquavella, MD, Principal Investigator, University of Rochester
Allocation: Not Applicable | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 35809
Record Dates: First submitted 2011-06-14; First posted 2011-06-17 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Dry Eye
Keywords: Dry Eye; tear film; lipid; tear volume; environmental chamber; thermal imaging
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drop Administration (Experimental)
  Interventions: Drug: B & L Soothe Lubricant Eye Drops; Drug: Liposic EDO; Drug: OcuFresh Eye Wash

INTERVENTIONS:
Drug: B & L Soothe Lubricant Eye Drops — Eye Drop
Drug: Liposic EDO — Eye Drop
Drug: OcuFresh Eye Wash — Saline drop

SUMMARY:
This study will evaluate ocular surface lubricants in subjects with dry eye syndrome.

DETAILED DESCRIPTION:
This study will objectively evaluate ocular surface lubricants in subjects with dry eye syndrome. Lubricants contain compounds that are purported to improve dry eye symptoms, although objective data is not available. The investigators seek to objectively evaluate the effectiveness of two lubricants and compare the results to a saline eye drop (control).

The investigators will assess the lipid layer before and after the administration of three products in the same eye of 25 dry eye subjects using the ellipsometry, imaging in a "normal" environment. Subsequently the investigators will change the environment to one that causes the subjects' ocular surface to experience "evaporative stress" (warmer, less humid and greater air flow) and perform the before and after drop administration measurements with the same three products in the same eye as the first environment.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-75 years
* Good general health
* Willing to spend time for the study; approximately one hour for a screening visit and 90 minutes for each of the measurement visits
* Currently using an OTC artificial tear for ocular comfort, at least occasionally.
* At least one positive dry eye symptom.

Exclusion Criteria:

* Current eye disease, infection or inflammation that requires the use of any prescription ocular medication.
* Recent past eye surgery.
* Female subjects may not be pregnant or lactating.
* Infectious diseases

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Tear Film Properties | Measurements: There is no time restriction between the screening and 1st measurement. 6 measurement visits occur approximately 7 days apart but can range from 3 to 14 days. The time between visit 3 and 4 are not be closer than 3 days, but no upper limit.
  The wavefront sensor instrument measures the eye's ability to create a sharp image.
  Ellipsometer (E) data identifies changes in lipid thickness and refractive index over the cornea.
  A thermal (T) imaging system provides thermal maps of the subject's eyes and face adjacent to the eyes.
  A questionnaire (Q) will ask subjects about their test eye's comfort. Subjects will be asked the questions prior to instillation of the eye drop and after each set of measurements.

CONTACTS AND LOCATIONS:
Overall Officials: James V Aquavella, MD, Principal Investigator — University of Rochester
Locations (1):
- Flaum Eye Institute at the University of Rochester, Rochester, New York, United States